CLINICAL TRIAL: NCT04817150
Title: LARC Study: Three-dimensional Versus Conventional 2D-laparoscopy for Rectocele and Rectal Prolapse Repair: a Prospective, Randomized, Single Center Study.
Brief Title: 3D vs 2D-laparoscopy for Rectocele and Rectal Prolapse Correction: a Prospective, Randomized, Single Center Study
Acronym: LARC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexander Khitaryan (Other)
Responsible Party: Sponsor-Investigator, Alexander Khitaryan, Professor, Private Healthcare Institution Clinical Hospital RGD-Medicine
Organization: Private Healthcare Institution Clinical Hospital RGD-Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LARC1
Record Dates: First submitted 2021-03-19; First posted 2021-03-26 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Rectocele; Female; Rectocele and Incomplete Uterine Prolapse; Rectocele and Complete Uterovaginal Prolapse; Rectal Prolapse
MeSH Terms: conditions — Rectocele; Prolapse; Rectal Prolapse

STUDY DESIGN:
Intervention Model Description: a prospective randomized comparative study in parallel groups
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes are assessed by 2 independent blinded coloproctologists
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-laparoscopy (Experimental): patients who underwent 3D laparoscopic ventral rectopexy
  Interventions: Procedure: Laparoscopic ventral mesh rectopexy
- 2D-laparoscopy (Active Comparator): patients who underwent conventional 2D laparoscopic ventral rectopexy
  Interventions: Procedure: Laparoscopic ventral mesh rectopexy

INTERVENTIONS:
Procedure: Laparoscopic ventral mesh rectopexy — Conventional laparoscopic ventral mesh rectopexy, as first described by D'Hoore

SUMMARY:
The aim is to compare proximate and remote results of 3D and conventional 2D laparoscopic interventions in terms of efficacy and safety in treatment of symptomatic rectocele and rectal prolapse.

This is a prospective randomized comparative study in parallel groups conducted in single Colorectal unit. Inclusion criteria: female patients with stage 3 rectocele (3-4 POP-Q [pelvic organ prolapse quantification] grade) and/or full-thickness rectal prolapse.

Intervention - laparoscopic ventral rectopexy. The primary outcome is objective cure rate of pelvic prolapse. Secondary outcomes include obstructive defecation and incontinence symptoms according to Wexner and Cleveland Clinic scales, and satisfaction according to Patient Global Impression of Improvement questionnaire. Operative times, intraoperative blood loss, length of hospital stay, postop pain severity, urinary incontinence, as well as surgical and mesh complications are also assessed.

The specific point of interest in this study is surgeon's tiredness after the operation assessed with Profile of Mood States questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* stage 3 rectocele (3-4 POP-Q grade) and/or full-thickness rectal prolapse
* age 18-70 y.o.

Exclusion Criteria:

* severe concomitants chronic diseases (American Society of Anesthesiologists class III - IV),
* ongoing oncological diseases,
* ongoing hematological diseases,
* ongoing inflammatory diseases of the colon and pelvic organs,
* pregnancy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
objective cure rate | 12 months postop
  objective cure rate according to clinical POP-Q assesment

SECONDARY OUTCOMES:
obstructive defecation cure | 12 months postop
  according to Wexner scale score (Cleveland Clinic Constipation Scoring System, scale of 0-30, with 0 = minimum, healthy individual and 30 = maximum, severe obstructive defecation)
incontinence cure | 12 months postop
  according to Cleveland Clinic scale score (Cleveland Clinic Incontinence Scoring System, scale of 0-20, with 0 = minimum, perfect continence and 20 = maximum, complete incontinence)
patient's satisfaction | 12 months postop
  according to PGII (Patient Global Impression of Improvement) questionnaire

OTHER OUTCOMES:
intraoperative blood loss | intraoperatively
  intraoperative blood loss (ml)
length of hospital stay | through study completion, an average of 1 year
  length of hospital stay (days)
postop pain severity | 24 hours postop
  VAS (Visual Analog Scale)
postop stress urinary incontinence | 12 months
  Valsalva test (positive - urinary incontinence presents, negative - no stress urinary incontinence)
complications rate | 12 months
  early and remote complications
surgeon's tiredness | 1 hour after the surgery
  Profile of Mood States Questionnaire
postoperative seroma/hematoma volume | 3 weeks
  size of liquid cavity surrounding mesh on 2-3 postoperative day and on 2-3 postoperative week (ml)
postop pain syndrom duration | through study completion, an average of 1 year
  pain medications consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Private Healthcare Institution Clinical Hospital "RGD-Medicine" Rostov-on-Don", Rostov-on-Don, Russia

IPD SHARING:
Plan to Share IPD: No